CLINICAL TRIAL: NCT03245528
Title: Expanded Access for LJPC-501
Status: Approved for marketing | Type: Expanded Access
Sponsor: La Jolla Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Other Study IDs: LJ501-EAP01
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Catecholamine Resistant Hypotension (CRH); Distributive Shock; High Output Shock; Sepsis; Vasodilatory Shock
MeSH Terms: conditions — Sepsis | interventions — Angiotensin I

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: LJPC-501 — angiotensin II

SUMMARY:
The primary objective of the study is to provide access to LJPC-501 for distributive shock patients who remain hypotensive despite receiving fluid and vasopressor therapy.

DETAILED DESCRIPTION:
Primary Objective

The primary objective of the study is to provide access to LJPC-501 for distributive shock patients who remain hypotensive despite receiving fluid and vasopressor therapy.

Secondary Objective

The secondary objective of the study is to assess the safety of LJPC-501.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be adults ≥ 18 years of age who remain hypotensive despite fluid therapy and vasopressor therapy and who received or are receiving a total sum norepinephrine (NE) equivalent unit dose of > 0.2 µg/kg/min for at least 2 hours prior to LJPC-501 infusion.
* Patients must have central venous access and an arterial line present, which is expected to remain for the duration of the LJPC-501 infusion.
* Patients must be adequately volume resuscitated in the opinion of the treating investigator.
* Patients must have clinical features of distributive shock documented by either estimated or measured CI > 2.3 L/min/m^2 determined by echocardiogram or another cardiac output monitoring modality OR a concurrent CVP > 8 mmHg and ScvO2 > 70%.
* Patient or legal surrogate is willing and able to provide informed consent per local guidance and patient/legal surrogate is willing to comply with all protocol requirements.

Exclusion Criteria:

* Patients with a MAP > 80 mmHg.
* Patients diagnosed with acute occlusive coronary syndrome requiring intervention.
* Patients who have been on ECMO < 6 hours.
* Patients in liver failure with a MELD score ≥ 30.
* Patients not mechanically ventilated with a history of asthma or who are currently experiencing bronchospasm requiring the use of inhaled bronchodilators.
* Patients with acute mesenteric ischemic or history of mesenteric ischemia.
* Patients with Raynaud's phenomenon, systemic sclerosis, or vasospastic disease.
* Patients with an expected lifespan of < 24 hours.
* Patients with active bleeding AND an anticipated need for transfusion of > 4 units PRBCs within 48 hours of the initiation of LJPC-501.
* Patients with active bleeding AND hemoglobin < 7 g/dL.
* Patients with an ANC < 500 cells/mm^3.
* Patients with a known allergy to mannitol.
* Patients who are currently participating in an investigational interventional trial.
* Women who are known to be pregnant at the time of Screening or have a positive serum or urine β-hCG, if of childbearing potential.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult